CLINICAL TRIAL: NCT01961362
Title: Observing the Effects of Supplemental Oxygen on Patients With Pulmonary Fibrosis
Brief Title: Supplemental Oxygen in Pulmonary Fibrosis
Status: Completed | Type: Observational
Sponsor: National Jewish Health (Other)
Collaborators: Pulmonary Fibrosis Foundation (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PCORI 4134a
Record Dates: First submitted 2013-10-09; First posted 2013-10-11 (Estimated); Results first posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Pulmonary Fibrosis
Keywords: Pulmonary fibrosis; Interstitial lung disease; Connective tissue disease; Chronic hypersensitivity pneumonitis; Idiopathic pulmonary fibrosis; Pulmonary fibrosis of any cause; Primary supporters/caregivers
MeSH Terms: conditions — Pulmonary Fibrosis; Lung Diseases, Interstitial; Connective Tissue Diseases; Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pulmonary fibrosis patients: Patients with pulmonary fibrosis of any cause (idiopathic, connective tissue disease, chronic hypersensitivity pneumonitis)

SUMMARY:
To enhance understanding of supplemental oxygen-its utility in and adoption by patients with pulmonary fibrosis-by examining how patients perceive it and by determining how perceptions and patient-centered outcome measures change from before to after supplemental oxygen is prescribed.

DETAILED DESCRIPTION:
The investigators aim to recruit patients with PF to participate in interviews and/or a one-year study of supplemental oxygen (O2). In the one-year study, the investigators will collect data before and for one year after PF patients are prescribed daily-use supplemental oxygen and compare outcomes, including shortness of breath, quality of life, fatigue, cough, and day-to-day functioning before and after O2.

ELIGIBILITY:
Inclusion Criteria:

Patient-Participants

(Using daily 02 therapy at time of enrollment)

* Diagnosis of PF
* Able to read and speak English
* Has been on daily-use supplemental oxygen for more than one year

(Not using daily 02 therapy at time of enrollment)

* Diagnosis of PF
* Able to read, speak and write in English
* Has not been prescribed daily-use supplemental oxygen
* Forced vital capacity <75% and diffusing capacity <65% of predicted values
* Subject's physician allows the subject to abstain from daily-use supplemental oxygen for 7-10 days after prescription to allow data for collection

Primary Supporters

* Self-report status of providing care or support to a person living with pulmonary fibrosis who has used supplemental oxygen for more than one year
* Able to speak English

O2 Prescribers

* Self-report status of being a prescriber of daily-use supplemental oxygen to PF patients
* Able to speak English

Exclusion Criteria:

Patient-Participants (Using daily 02 therapy at time of enrollment)

* No diagnosis of PF
* Unable to read and speak English
* Has been on daily-use supplemental oxygen for less than one year

(Not using daily 02 therapy at time of enrollment)

* No diagnosis of PF
* Unable to read, speak and write in English
* Using supplemental oxygen during the day
* Subject's physician does not allow the subject to abstain from daily-use supplemental oxygen for 7-10 days after prescription to allow data for collection

Primary Supporters • Not meeting inclusion criteria

O2 Prescribers

• Not meeting inclusion criteria

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with pulmonary fibrosis of any cause (idiopathic, related to connective tissue disease [e.g., rheumatoid arthritis, systemic sclerosis/scleroderma, dermato-/polymyositis, sjogren's syndrome], familial or genetic) or the primary supporter/caregiver of a patient with pulmonary fibrosis
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2013-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Swigris, DO, MS, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health Interstitial Lung Disease Program, Denver, Colorado, United States

REFERENCES:
- [Derived] Root ED, Graney B, Baird S, Churney T, Fier K, Korn M, McCormic M, Sprunger D, Vierzba T, Wamboldt FS, Swigris JJ. Physical activity and activity space in patients with pulmonary fibrosis not prescribed supplemental oxygen. BMC Pulm Med. 2017 Nov 23;17(1):154. doi: 10.1186/s12890-017-0495-2. PMID 29169394
- [Derived] Olson AL, Graney B, Baird S, Churney T, Fier K, Korn M, McCormick M, Sprunger D, Vierzba T, Wamboldt FS, Swigris JJ. Tracking dyspnea up to supplemental oxygen prescription among patients with pulmonary fibrosis. BMC Pulm Med. 2017 Nov 22;17(1):152. doi: 10.1186/s12890-017-0497-0. PMID 29166901
- [Derived] Graney BA, Wamboldt FS, Baird S, Churney T, Fier K, Korn M, McCormick M, Vierzba T, Swigris JJ. Informal caregivers experience of supplemental oxygen in pulmonary fibrosis. Health Qual Life Outcomes. 2017 Jul 1;15(1):133. doi: 10.1186/s12955-017-0710-0. PMID 28668090

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We enrolled patients with PF not using supplemental O2 and then followed them forward until they were prescribed supplemental O2 by their treating practitioner, and then we followed them for an additional 12 months after being prescribed O2.
Pre-assignment Details: We enrolled 19 subjects.
Period: Overall Study
Arm/Group | Pulmonary Fibrosis Patients
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: We enrolled patients with PF not using supplemental O2 and then followed them forward until they were prescribed supplemental O2 by their treating practitioner, and then we followed them for an additional 12 months after being prescribed O2.
Groups:
- Pulmonary Fibrosis Patients: Patients with pulmonary fibrosis of any cause (idiopathic, connective tissue disease, chronic hypersensitivity pneumonitis). We enrolled patients with PF not using supplemental O2 and then followed them forward until they were prescribed supplemental O2 by their treating practitioner, and then we followed them for an additional 12 months after being prescribed O2.
Arm/Group | Pulmonary Fibrosis Patients
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants] — Age of the subjects
  Participants
    <=18 years | 0
    Between 18 and 65 years | 7
    >=65 years | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 19
Percentage of Predicted Forced Vital Capacity [Mean (Standard Deviation); unit: Percentage of predicted FVC] | 64.9 (16.1)
University of California San Diego Shortness of Breath Questionnaire [Mean (Standard Deviation); unit: units on a scale] — The University of California San Diego Shortness of Breath Questionnaire (or UCSD SOB) is a tool that measures shortness of breath using 24 items, each with response options ranging from 0 to 5, corresponding to "None at all" and "Maximally or unable to do because of breathlessness." Thus, scores for the UCSD SOB range from 0 to 120, with higher scores indicating greater shortness of breath.
  units on a scale | 32.9 (14.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in University of California San Diego Shortness of Breath Questionnaire From Immediately Prior to One Month After Starting Daily-use Supplemental Oxygen
Description: The University of California San Diego Shortness of Breath Questionnaire (or UCSD SOB) is a tool that measures shortness of breath using 24 items, each with response options ranging from 0 to 5, corresponding to "None at all" and "Maximally or unable to do because of breathlessness." Thus, scores for the UCSD SOB range from 0 to 120, with higher scores indicating greater shortness of breath.
Time Frame: UCSD SOB score at one month after being prescribed supplemental O2
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Pulmonary Fibrosis Patients
Number analyzed (Participants) | 19
points | 0.9 (8.7)
Statistical Analysis 1: Comparison: Pulmonary Fibrosis Patients; Test type: Superiority; p = 0.6, t-test, 2 sided — P<0.05 considered to represent statistical significance; Mean Difference (Net) = 0.9, Standard Deviation 0.87
Statistical Analysis 2: Comparison: Pulmonary Fibrosis Patients; Test type: Superiority; p < 0.05, Mixed Models Analysis; Mean Difference (Net) = -0.07, Standard Error of Mean 1.2

2. Secondary Outcome: Change in Physical Component Summary (PCS) Score From the Medical Outcomes Study Short-Form, 36-item Questionnaire (SF-36).
Description: The PCS of the SF-36 assesses a domain of quality of life. Its scores range from 0-100, with higher scores indicating better quality of life on this domain.
Time Frame: One month after daily-use supplemental oxygen implementation
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Pulmonary Fibrosis Patients
Number analyzed (Participants) | 19
units on a scale | -0.07 (1.2)
Statistical Analysis 1: Comparison: Pulmonary Fibrosis Patients; Test type: Superiority; p < 0.05, Mixed Models Analysis; Median Difference (Net) = -0.07, Standard Error of Mean 1.2

3. Secondary Outcome: Fatigue Severity Scale
Description: The Fatigue Severity Scale is a 9-item questionnaire, scored from 9-63, with higher scores indicating more severe fatigue.
Time Frame: One month after daily-use supplemental oxygen implementation
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Pulmonary Fibrosis Patients
Number analyzed (Participants) | 19
units on a scale | 5.2 (2.4)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Pulmonary Fibrosis Patients
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

LIMITATIONS AND CAVEATS:
Fewer patients than expected were prescribed supplemental O2 by their practitioners; thus, our study was under-powered for the primary and secondary outcome assessments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No